CLINICAL TRIAL: NCT07126379
Title: The Family Foundations Trial: Promoting Family Wellbeing in Regional and Rural Communities Affected by Environmental Threats
Brief Title: The Family Foundations Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deakin University (Other)
Collaborators: La Trobe University (Other); Holstep Health (Unknown); Colac Area Health (Unknown); Brophy Family & Youth Service (Unknown); The Bridge (Unknown); Kids First (Unknown); Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117878
Record Dates: First submitted 2025-08-08; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Outcomes
Keywords: mental health; parent mental health; coparenting; rural health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a parallel group multi-site randomised controlled trial. FF (8 session family-based intervention) will be compared to a brief intervention (single brief telephone consultation + resources + referral). FF will be delivered via telehealth from 5 rural health service sites. Families (comprised of at least two parents/caregivers) will be randomised in a 1:1 ratio to the two treatment arms. The trial is open label.
  This trial will be registered within the Australian Teletrial Program. A teletrial is a group of clinical Satellite Sites working together to conduct a clinical trial, consisting of a Primary Site (Deakin; assuming overall responsibility for the conduct of the trial) and 5 Satellite Sites who will deliver the FF intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Foundations (Experimental): Families allocated to FF will receive the program via one of the trial satellite sites within 2 weeks of randomisation.
  Interventions: Behavioral: Family Foundations
- Family Life Check In (Active Comparator): Families allocated to the Family Life Check-In will receive this condition from a Clinical Research Nurse, employed through the primary site (Deakin University) within 2 weeks of randomisation.
  Interventions: Behavioral: Family Life Check-In

INTERVENTIONS:
Behavioral: Family Foundations — FF is an 8-session program for families of children aged 0-12 years targeting parent mental health and family conflict. It will be delivered via telehealth by an allied health professional (i.e., social work, psychology, counselling qualification) trained in FF. The 8 sessions can be delivered flexibly (1 or 2 sessions per week). The duration between sessions can vary as per the needs of the family. We are allowing up to 11 weeks from randomisation for FF to be completed. FF is a manualised program which provides instruction on discussion activities, skills practice, video and workbook exercises for every session. Sessions are based around the content areas of: emotion regulation, stress management, healthy communication, coparenting, conflict resolution, and problem solving.
  Arms: Family Foundations
Behavioral: Family Life Check-In — Families allocated to Family Life Check In will receive this condition from a Clinical Research Nurse, employed at the Primary site (deakin University) with 2 weeks of randomisation. This brief intervention will be comparable to care typically provided to parents/caregivers seeking support for mental health difficulties and/or family/parent relationships issues from a community health service at intake. Family Life Check-In involves a brief (~30 minute) telephone consultation involving: a) an assessment of the families' needs with one or all parents, b) referral to local services including GP to discuss a mental health care plan, c) provision of reputable Australian web-based resources about supporting children during crises (Raising Children Network, Phoenix Disaster Recovery), and (d) telephone and online support services (BeyondBlue; Lifeline, PANDA, MensLine, KidsLine, Parentline).
  Arms: Family Life Check In

SUMMARY:
In this project, researchers are exploring different ways to support the wellbeing and relationships of families with young children (0-12 years). People in regional and rural communities often live with the threat of bushfires, floods, drought, severe storms, and other extreme weather events. Some families have been affected by these disasters and are still trying to recover.

Researchers will test two different ways of supporting families in regional and rural Victoria:

Family Foundations (FF): An 8-session program to promote parent wellbeing, parenting partnerships, and communication. All parents/caregivers/parenting partners in the family participate in sessions delivered by a health professional online.

Family Life Check-In: A brief 30-minute telephone call with a health professional to discuss family wellbeing and relationships, and identify any supports needed.

The goal of this trial is to learn whether FF works to reduce mental health difficulties for regional and rural families. The main question it aims to answer is:

Compared to Family Life Check-In, does Family Foundations lead to fewer mental health difficulties?

Participants will:

Complete an online survey before randomisation, after they have received FF or Family Life Check-In, and six months after starting the project.

Take part in either Family Foundations or Family Life Check-In.

DETAILED DESCRIPTION:
Study Design This is a parallel-group, multi-site, randomised controlled trial. Family Foundations (FF), an 8-session family-based intervention, will be compared to a brief intervention (single brief telephone consultation plus resources and referral). FF will be delivered via telehealth from five rural health service sites. Families (comprised of at least two parents/caregivers) will be randomised in a 1:1 ratio to the two treatment arms. The trial is open-label.

This trial will be registered within the Australian Teletrial Program. A teletrial is a group of clinical satellite sites working together to conduct a clinical trial, consisting of a Primary Site (Deakin University, which assumes overall responsibility for the conduct of the trial) and five satellite sites that will deliver the FF intervention. These sites are: Holstep Health, Kids First, Colac Area Health, The Bridge Youth Service, and Brophy Family and Youth Service.

Study Aims

There are two main aims of this study:

Aim 1: To evaluate the effectiveness of FF in reducing mental health difficulties for rural families.

We hypothesise that, compared to a brief intervention (single telephone consultation plus resources and referral), FF will lead to fewer parent mental health difficulties (primary outcome at 24 weeks post-randomisation).

Aim 2: To assess the implementation of FF and the brief intervention, including:

1. Reach and uptake of FF by rural families
2. Experiences of care for families receiving FF or the brief intervention
3. Intervention fidelity
4. Enablers and barriers to implementation and adoption (not covered in this protocol)
5. Workforce knowledge, skills, and confidence to provide mental health care to families (not covered in this protocol)

Participants Participants will be 236 families (at least 472 parents/caregivers) of children aged 0-12 years, living in regional or rural areas of Australia. At least two parents/caregivers in each family must agree to participate, as this is a family intervention, but they are not required to be in a couple relationship or living together.

Recruitment Families living in regional and rural areas will be invited to participate in a study about ways to promote and protect the wellbeing of families in country Australia, particularly those currently or recently (within the past five years) experiencing environmental threats (e.g., drought, floods, severe storms, bushfires).

Study promotion and recruitment will occur across a range of settings, including the general public, community services, and through our partners (Royal Flying Doctor Service - Victoria; National Centre for Farmer Health). Recruitment strategies, co-designed with our partners and lived-experience group, will include a mix of active and passive approaches.

Intervention Arms The FF program (intervention) will be compared to the brief intervention (control), referred to as Family Life Check-In. This name will be used consistently in all study materials and in the PICF.

Families allocated to FF will receive the program via one of the trial satellite sites within two weeks of randomisation. Satellite sites will indicate their capacity to deliver FF to allocated families regardless of the family's location.

FF is an 8-session, manualised program for families of children aged 0-12 years, targeting parent mental health and family conflict. It is delivered via telehealth by allied health professionals (e.g., social workers, psychologists, or counsellors) trained in FF. Sessions may be delivered flexibly (1-2 per week), with up to 11 weeks allowed from randomisation to completion. Each session includes discussion activities, skills practice, videos, and workbook exercises. Content areas include emotion regulation, stress management, healthy communication, co-parenting, conflict resolution, and problem-solving.

Families allocated to the brief intervention will receive support from a Clinical Research Nurse employed at the primary site (Deakin University), who is a qualified maternal and child health nurse with experience supporting parents and families. Within two weeks of randomisation, the nurse will conduct a brief (~30-minute) telephone consultation that includes:

1. Assessment of family needs with one or more parents
2. Referral to local services, including a GP to discuss a mental health care plan
3. Provision of reputable Australian web-based resources (e.g., Raising Children Network, Phoenix Disaster Recovery)
4. Referral to telephone/online support services (e.g., Beyond Blue, Lifeline, PANDA, MensLine, Kids Helpline, Parentline)

Data Collection

Participants will complete online self-report surveys at three time points:

Baseline (~2 weeks prior to randomisation)

12 weeks after randomisation

24 weeks after randomisation

Participants will also be invited to a qualitative interview at 24 weeks. Details of the outcome measures are provided in the uploaded study protocol and the 'Outcome Measures' section of this form.

Data Analysis A detailed statistical analysis plan will be prepared by Dr Anneke Grobler before database lock. Analyses will follow the intention-to-treat (ITT) principle. Continuous endpoints (primary and secondary outcomes) will be analysed using linear regression, adjusting for treatment arm, health service site, and baseline scores. Clustering at the family level will be accounted for using appropriate statistical models.

Mean differences between treatment arms will be reported with 95% confidence intervals. Risk differences will be calculated using a generalised linear model (GLM) with an identity link function and binomial family, including treatment arm, health service site, and baseline scores. Standard errors will be clustered at the family level.

Health Economic Analysis Health economic analysis will be led by Professor Suzanne Robinson at Deakin University. A cost-consequences analysis will present the incremental cost of the intervention (intervention plus service use) minus control group costs, alongside all outcome measures. A cost-effectiveness analysis will estimate the incremental cost per: Unit reduction in distress score (K6 or DASS-21); QALY gained (via AQoL-8D).Results will be reported in line with CHEERS guidelines. A modelled estimate of costs and cost-effectiveness for scale-up will be developed in collaboration with service partners, based on current capacity and anticipated need. Sensitivity analyses will assess the robustness of findings.

Dissemination and Translation Plan Findings will be reported to the Medical Research Future Fund: Million Minds Mission (MRFF) through progress and final reports. Results will also be disseminated via conference presentations and at least two peer-reviewed publications. Only aggregated, de-identified group data will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Family must be living in a regional or rural area
* Family must have at least one child aged 0-12 years
* At least 2 parents/caregivers in the family must agree to participate in evaluation, and FF, if allocated. (Please note: A family member or someone else involved in raising children in the family may participate in FF. Families are not required to be in a couple relationship or living together).
* At least one parent/caregiver within the family reports mental health difficulties and/or two or more risk factors for poor mental health in the last 5 years including (a) experienced a recent or past natural disaster (i.e., drought, flood, fire, severe storm), (b) living with the threat of a natural disaster (i.e., bushfires during summer), (c) self-reported history of poor mental health, (d) financial hardship, (e) young parental age at time of first baby (18-25yrs), (f) relationship conflict, or (g) social isolation.

Exclusion Criteria:

* At least one parent has a severe mental health disorder - self reported psychosis, substance use dependency, prescribed anti-psychotic medication that may interfere with their ability to take part in the trial and in the FF intervention if allocated. They may require more intensive mental health interventions and treatment than what can be provided by the trial interventions.
* The family has an overt indicator of family violence - self-reported intervention order or court case for family violence.
* The family has child protection service involvement - self-reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Mental Health Difficulties. The Depression Anxiety Stress Scale-21 (DASS-21), mean difference in total scale scores between FF and Usual Care arms | 24-weeks post-randomisation
  The Depression Anxiety Stress Scale-21 (DASS-21) assesses symptoms of depression, anxiety, and stress in the past week (21 items). The items are rated on a 4-point scale ranging from 0-Never to 3-Almost Always. A total scale score can be created, as well as specific subscales for depressive, anxiety and stress symptoms. Higher scores indicate greater levels of mental health difficulties. Excellent reliability and validity has been demonstrated in Australian population-based samples. The DASS-21 is routinely used by early parenting services.

SECONDARY OUTCOMES:
Mental Health Difficulties. The Depression Anxiety Stress Scale-21 (DASS-21), mean difference in total scale and subscale scores between FF and Usual Care arms | 12-weeks post-randomisation
  The Depression Anxiety Stress Scale-21 (DASS-21) assesses symptoms of depression, anxiety, and stress in the past week (21 items). The items are rated on a 4-point scale ranging from 0-Never to 3-Almost Always. A total scale score can be created, as well as specific subscales for depressive, anxiety and stress symptoms. Higher scores indicate greater levels of mental health difficulties. Excellent reliability and validity has been demonstrated in Australian population-based samples. The DASS-21 is routinely used by early parenting services.
Mental Health Difficulties. The Depression Anxiety Stress Scale-21 (DASS-21), mean difference in subscale scores between FF and Usual Care arms | 24-weeks post-randomisation
  The Depression Anxiety Stress Scale-21 (DASS-21) assesses symptoms of depression, anxiety, and stress in the past week (21 items). Scores on each scale range from 0-42 with higher scores indicating a greater severity of symptoms. Clinical ranges are available. Excellent reliability and validity has been demonstrated in Australian population-based samples. The DASS-21 is routinely used by early parenting services.
Kessler Psychological Distress Scale - 6, mean difference in total score between the Family Foundations and Usual Care arms. | 12-weeks post-randomisation
  The 6-item Kessler Psychological Distress Scale (K6) assesses general symptoms of depression and anxiety in the last 30 days/4 weeks. The 6 items are rated on a 5-point scale ranging from 0-None of the time to 4-All of the time. Higher scores indicate higher levels of psychological distress. The K6 is widely used in clinical trials for common mental health disorders, and is consistent with a transdiagnostic approach proposing a common set of psychological distress symptoms underlie mood and anxiety disorders . It has well-established symptomatic and clinical cut-points, high specificity (0.96), robust total classification accuracy (0.92) to identify mood and anxiety disorders [32], and correlates with validated measures of suicidality [45]. Australian population data for men are available using the K6 (e.g. National Survey of Mental Health and Wellbeing, Longitudinal Study of Australian Children). The study investigators have published extensively on fathers' mental health.
Kessler Psychological Distress Scale- 6, mean difference in total score between the Family Foundations and Usual Care arms. | 24-weeks post-randomisation
  The 6-item Kessler Psychological Distress Scale (K6) assesses general symptoms of depression and anxiety in the last 30 days/4 weeks. The 6 items are rated on a 5-point scale ranging from 0-None of the time to 4-All of the time. Higher scores indicate higher levels of psychological distress. The K6 is widely used in clinical trials for common mental health disorders, and is consistent with a transdiagnostic approach proposing a common set of psychological distress symptoms underlie mood and anxiety disorders . It has well-established symptomatic and clinical cut-points, high specificity (0.96), robust total classification accuracy (0.92) to identify mood and anxiety disorders [32], and correlates with validated measures of suicidality [45]. Australian population data for men are available using the K6 (e.g. National Survey of Mental Health and Wellbeing, Longitudinal Study of Australian Children). The study investigators have published extensively on fathers' mental health.
Parental conflict. The Communication and Problem Solving Scale, mean difference in subscale scores between the Family Foundations and the Usual Care arms. | 12 weeks post-randomisation
  The Communication and Problem Solving Scale consists of 35 items and asks parents about a broad range of behaviours (e.g., 'talk it out with one another; change the subject; threaten to end the relationship) when having a disagreement with their co-parent. Items are rated on a 4-point scale from 1 = Never to 4 = Often. There are six subscales assessing Cooperation, Avoidance, Child Involvement, Stalemating, Verbal Aggression and Physical Aggression. Subscale and total scale scores can be computed with higher scores indicating more frequent engagement in conflict behaviours. The scale has established reliability and validity, and has been used in evaluations of FF in Australia.
Parental conflict. The Communication and Problem Solving Scale , mean difference in subscale scores between the Family Foundations and the Usual Care arms. | 24 weeks post-randomisation
  The Communication and Problem Solving Scale consists of 35 items and asks parents about a broad range of behaviours (e.g., 'talk it out with one another; change the subject; threaten to end the relationship) when having a disagreement with their co-parent. Items are rated on a 4-point scale from 1 = Never to 4 = Often. There are six subscales assessing Cooperation, Avoidance, Child Involvement, Stalemating, Verbal Aggression and Physical Aggression. Subscale and total scale scores can be computed with higher scores indicating more frequent engagement in conflict behaviours. The scale has established reliability and validity, and has been used in evaluations of FF in Australia.
Co-parenting. The Coparenting Relationship Scale, mean difference in subscale scores between FF and the brief intervention arms. | 12-weeks post randomisation
  The Coparenting Relationship Scale consists of 35 items (e.g., my co-parent asks my opinion on issues related to parenting, my co-parent has lots of patience with our child, my relationship with my co-parent is stronger now than before we had a child), comprising seven subscales (Coparenting Agreement, Coparenting Closesness, Exposure to Conflict, Coparenting Support, Coparenting Undermining, Endorse Co-parent Parenting, and Division of Labor). Each item is rated on a 7-point scale, ranging from 0=Not true of us/Never to 6=Very true of us/Often. Particular items are reverse scored, and then summed. The scale is ideal for examining the role of coparenting in diverse family contexts. The subscales have excellent internal reliability with parent populations in the US and Australia.
Co-parenting. The Coparenting Relationship Scale, mean difference in subscale scores between FF and the brief intervention arms. | 24-weeks post randomisation
  The Coparenting Relationship Scale consists of 35 items (e.g., my co-parent asks my opinion on issues related to parenting, my co-parent has lots of patience with our child, my relationship with my co-parent is stronger now than before we had a child), comprising seven subscales (Coparenting Agreement, Coparenting Closesness, Exposure to Conflict, Coparenting Support, Coparenting Undermining, Endorse Co-parent Parenting, and Division of Labor). Each item is rated on a 7-point scale, ranging from 0=Not true of us/Never to 6=Very true of us/Often. Particular items are reverse scored, and then summed. The scale is ideal for examining the role of coparenting in diverse family contexts. The subscales have excellent internal reliability with parent populations in the US and Australia.
Anger. Dimensions of Anger Reactions (DAR-5), The mean difference in DAR-5 between FF and brief intervention arms. | 24-weeks post randomisation
  The Dimension of Anger Reactions (DAR-5) is a 5-item self- measure of experiences of anger which assesses the frequency, intensity, duration, aggression and impact on a person's social functioning over the past 4-weeks. Items are rated on a 5-point scale, ranging from 1 = None or almost none of the time to 5 = All or almost all of the time, where higher scores indicate worse symptomology, and a score greater than 12 indicated problem anger.
Wellbeing. Warwick Edinburgh Mental Wellbeing Scale Short form (SWEMWBS), mean difference in wellbeing between the FF and brief intervention arms. | 12-weeks post randomisation
  To focus on the positive aspects of mental health, the Warwick Edinburgh Mental Wellbeing Scale Short form (SWEMWBS) will be used to assess thoughts and feelings which relate to mental wellbeing. The 7-items assessing a range of positive thoughts and experiences related to mental health (e.g., I have been feeling optimistic about the future; I've been dealing with problems well; I have been thinking clearly) in the last 2 weeks on a 5-point scale from 1 = None of the time to 5 = All of the time. Items scores were summed, with higher scores indicating higher overall wellbeing.
Wellbeing. Warwick Edinburgh Mental Wellbeing Scale Short form (SWEMWBS), mean difference in wellbeing between the FF and brief intervention arms. | 24-weeks post randomisation
  To focus on the positive aspects of mental health, the Warwick Edinburgh Mental Wellbeing Scale Short form (SWEMWBS) will be used to assess thoughts and feelings which relate to mental wellbeing. The 7-items assessing a range of positive thoughts and experiences related to mental health (e.g., I have been feeling optimistic about the future; I've been dealing with problems well; I have been thinking clearly) in the last 2 weeks on a 5-point scale from 1 = None of the time to 5 = All of the time. Items scores were summed, with higher scores indicating higher overall wellbeing.
Child-Parent Relationship. Child-Parent Relationship Scale-short form (CPRS), mean difference in the conflict and closeness subscale scores between the FF and brief intervention arms. | 24-weeks post randomisation
  The Child-Parent Relationship Scale- short form (CPRS) assesses parents' perceptions of their relationship with their child. The scale consists of 15-items that assess parents' perceptions of their relationship with their child (e.g., 'I share an affectionate, warm relationship with my child'). Items were rated on a 5-point scale ranging from 1= definitely does not apply to 5 = definitely applies. There are two subscales assessing (1) Closeness and (2) Conflict. Item scores were summed with higher scores indicating higher closeness or conflict in the parent-child relationship.
Parenting hostility. The Brief Co-parental Communication Scale , The mean difference in parenting hostility scores between the FF and brief intervention arms. | 24-weeks post randomisation
  The brief Co-parental Communication Scale used in the Longitudinal Study of Australian Children which consists of five items assessing how often parents engage in verbal conflict (e.g. 'How often do you argue?') and one item assessing how often they engage in physical conflict (e.g. 'How often do you have arguments with your co-parent that end up with people pushing, hitting, kicking or shoving?'). The items are rated on a 5-point scale from 1 = never to 5 = always. Items scores were summed, with higher scores indicating more frequent interparental conflict. The scale has excellent reliability and validity in Australian populations.
Quality of life. The Assessment of Quality of Life 8 dimension (AQoL-8D), mean difference in quality of life subscales scores between the FF and brief intervention arms. | 24-weeks post randomisation
  The Assessment of Quality of Life 8 dimension (AQoL-8D). It is a validated tool assessing quality of life impacts in the economic evaluation. Australian population normative data are available and will be used to determine preference weighted health related quality of life utility scores ranging from 0-1 with higher scores indicating higher quality of life. The AQoL-8D is particularly suited to measuring mental health aspects of quality of life. Participants will complete the scale via an online REDCap survey.
Traumatic Stress Symptoms. The Brief PTSD Checklist, the difference in proportion of participants meeting the clinical cut off between the FF and usual care will be assessed. | 24-weeks post randomisation
  The brief version of the PTSD Checklist is a self-report 4-item screening tool for the presence of trauma symptoms in the last 4 weeks. The measures asks participants to rate the extent to which they have experienced four diagnostic symptoms of PTSD in the past month. Participants are asked to rate the extent that they are bothered by a traumatic event on a 5 point scale (0 = not at all to 4 = Extremely).
Suicidal Ideation. The Suicidal Ideation Attributes Scale (SIAS), risk difference between FF and the brief intervention arms. | 12-weeks post randomisation
  Suicidal ideation will be assessed using the Suicidal Ideation Attributes Scale (SIAS). The SIAS is a self-reported 5-item screening tool for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Any ideation is indicative of risk for suicidal behaviour (scores >1 indicate risk).
Suicidal Ideation. The Suicidal Ideation Attributes Scale (SIAS), risk difference between FF and the brief intervention arms. | 24-weeks post randomisation
  Suicidal ideation will be assessed using the Suicidal Ideation Attributes Scale (SIAS). The SIAS is a self-reported 5-item screening tool for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Any ideation is indicative of risk for suicidal behaviour (scores >1 indicate risk).
Suicidal Ideation. The Suicidal Ideation Attributes Scale (SIAS), mean difference in total scale score between FF and the brief intervention arms. | 12-weeks post randomisation
  Suicidal ideation will be assessed using the Suicidal Ideation Attributes Scale (SIAS). The SIAS is a self-reported 5-item screening tool for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Any ideation is indicative of risk for suicidal behaviour (scores >1 indicate risk).
Suicidal Ideation. The Suicidal Ideation Attributes Scale (SIAS), mean difference in total scale score between FF and the brief intervention arms. | 24-weeks post randomisation
  Suicidal ideation will be assessed using the Suicidal Ideation Attributes Scale (SIAS). The SIAS is a self-reported 5-item screening tool for the presence and severity of suicidal thoughts in the last month based on frequency, controllability, closeness to attempt, level of distress, and impact on daily functioning. Any ideation is indicative of risk for suicidal behaviour (scores >1 indicate risk).
Health Service Use cost, mean difference in cost of healthcare use between the FF and Usual Care arms | 24-Weeks post randomisation
  Health dervice use will be assessed by self-reported type and costof healthcare services accessed (prior to baseline and during the study period).
Health Service Use, mean difference in number of healthcare use between the FF and Usual Care arms | 24-Weeks post randomisation
  Health dervice use will be assessed by self-reported type and number healthcare services accessed (prior to baseline and during the study period).
Productivity. The Work Productivity and Activity Impairment Questionnaire: General Health (WPAI), mean difference in total scores between the FF and Usual Care arms | 24-weeks post randomisation
  the Work Productivity and Activity Impairment Questionnaire: General Health (WPAI) which is a measure of impairments in both paid and unpaid work. Participants are asked 6-items (e.g., are you currently employed, hours missed due to a health problem, hours worked and degree health has affected productivity while at work on a Visual Analogue Scale) for the past seven days. It is well validated among specific health problems and between clinical treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Giallo, Principal Investigator — Deakin University
Locations (6):
- Australia (6):
  - Deakin University, Burwood, Victoria
  - Colac Area Health, Colac, Victoria
  - Holstep Health, Melbourne, Victoria
  - The Bridge Youth Service, Shepparton, Victoria
  - Kids First, Wallan, Victoria
  - Brophy Family & Youth Services, Warrnambool, Victoria

IPD SHARING:
Plan to Share IPD: No
We will not seek consent from participants to share their data, and we do not have ethics approval to share individual participant data.